CLINICAL TRIAL: NCT06025396
Title: A Phase 1, Randomized, Placebo-Controlled, Multiple Ascending Dose (MAD) Study To Evaluate The Safety, Tolerability, and Pharmacokinetics of TMP-301 in Healthy Subjects
Brief Title: Multiple Ascending Dose Study of TMP-301 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tempero Bio, Inc. (Industry)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: TMP-301-HNV-101; U01DA057118 (NIH)
Record Dates: First submitted 2023-08-21; First posted 2023-09-06 (Actual); Results first posted 2025-07-29 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Cocaine Use Disorder; Substance Use Disorders; Healthy Volunteers
Keywords: drug addiction; cocaine use disorder; cocaine dependance; TMP-301; cocaine use; CUD; drug abuse
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Intervention Model Description: sequential assignment
Who Masked: Participant, Investigator
Masking Description: Double blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Active TMP-301 (Experimental): Cohort 1= 50mg, capsules form, one capsule - two times per day - total 100mg/day;
  Cohort 2= 50mg, capsule form, 1 capsules - one time per day- total 50mg/day
  Cohort 3= 50mg, capsule form, 2 capsules - one time per day- total 100mg/day;
  Cohort 4 = Dose Titration: 50mg, capsule form, 1 capsules - one time per day - total 50 mg/day - on Days 1-7; and 50 mg, capsule form, 2 capsules - one time per day - total 100mg/day - on Days 8-14;
  Each cohort duration is 14 days of dosing
  Interventions: Drug: Cohort 1 - TMP-301; Drug: Cohort 2 - TMP-301; Drug: Cohort 3 - TMP-301; Drug: Cohort 4 - TMP-301
- Placebo (Placebo Comparator): Cohort 1= Placebo, capsules form, one capsule - two times per day;
  Cohort 2= Placebo, capsule form, 1 capsules - one time per day;
  Cohort 3= Placebo, capsule form, 2 capsules - one time per day;
  Cohort 4 = Dose Titration: Placebo, capsule form, 1 capsules - one time per day - on Days 1-7; and Placebo, capsule form, 2 capsules - one time per day - on Days 8-14;
  Each cohort duration is 14 days of dosing
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cohort 1 - TMP-301 — 50 mg BID Fasted
  Arms: Active TMP-301
Drug: Placebo — Multiple ascending dose comparator
  Arms: Placebo
Drug: Cohort 2 - TMP-301 — 50 mg QD Fasted
  Arms: Active TMP-301
Drug: Cohort 3 - TMP-301 — 50 mg QD Fed
  Arms: Active TMP-301
Drug: Cohort 4 - TMP-301 — 25 mg QD Fed
  Arms: Active TMP-301

SUMMARY:
A PHASE 1, RANDOMIZED, PLACEBO CONTROLLED, MULTIPLE ASCENDING DOSE (MAD) STUDY TO EVALUATE THE SAFETY, TOLERABILITY, AND PHARMACOKINETICS OF TMP-301 IN HEALTHY SUBJECTS.

DETAILED DESCRIPTION:
This study will be a randomized, double-blind, placebo controlled, fixed sequence, MAD study. The study will be conducted in a single clinical research unit (CRU). The study will consist of up to 4 cohorts. Subjects will only participate in 1 cohort.

Screening will occur within approximately 28 days prior to the first scheduled study drug administration. Subjects who meet all inclusion criteria and none of the exclusion criteria and who consent to participation will be admitted to the CRU for baseline evaluations prior to dosing.

Subjects will be fasted overnight for 10 hours prior to the morning dose, followed by a 2 hour fast. Subjects are fasted for 2 hours prior to dosing and 2 hours following the evening dose for the cohort 1 (50 mg bid).

Subjects will be discharged from the CRU on Day 18. Subjects will return to the CRU on Day 25 for a follow-up visit and EOS procedures.

Caffeine (100 mg) will be included as probe CYP1A2 substrate in cohort 2 and subsequent cohorts.

The maximum duration of subject participation, including Screening, will be approximately 53 days.

Subjects who terminate the study early will perform follow-up procedures at the time of Early Termination.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form (ICF)
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Healthy adult male or female
4. If male, meets one of the following criteria: a) Is able to procreate and agrees to use one of the accepted contraceptive regimens and not to donate sperm from the first study drug administration to at least 90 days after the follow-up visit. An acceptable method of contraception includes one of the following: Abstinence from heterosexual intercourse, or Male condom with spermicide or male condom with a vaginal spermicide (gel, foam, or suppository); or b) Is unable to procreate; defined as surgically sterile (ie, has undergone a vasectomy at least 180 days prior to the first study drug administration)
5. If female, meets one of the following criteria: (1) Physiological postmenopausal status, defined as the following: a) absence of menses for at least 12 months prior to the first study drug administration (without an alternative medical condition); and b) Follicle stimulating hormone (FSH) levels ≥ 40 mIU/mL at Screening; Or (2) Surgical postmenopausal status, defined as the following: a) bilateral oophorectomy, salpingectomy, or tubal ligation; hysterectomy
6. Aged at least 18 years but not older than 59 years, inclusive, at the time of informed consent
7. Body mass index (BMI) within 18.5 kg/m2 to 32.0 kg/m2, inclusively
8. Minimum body weight of at least 50.0 kg
9. Non- or ex smoker (An ex smoker is defined as someone who completely stopped using nicotine products for at least 90 days prior to the first study drug administration)
10. Must be willing to abstain from drinking coffee or caffeine containing beverages during the study, except where part of the study procedures
11. Has supine blood pressure and pulse rate within the following ranges after 5 minutes rest: systolic blood pressure 90 to 140 mmHg, diastolic blood pressure 50 to 90 mmHg, and pulse rate 45 to 90 bpm at Screening and on Day -1
12. Have no clinically significant diseases captured in the medical history or evidence of clinically significant findings on the physical examination (including vital signs) and/or ECG, as determined by an Investigator
13. Has clinical laboratory test results within the reference ranges of the testing laboratory, with the exception of results outside the reference ranges that are deemed not clinically significant by the Investigator (or designee) at Screening and check-in *

Exclusion Criteria:

1. Female who is lactating
2. Female who is pregnant according to the pregnancy test at Screening or prior to the first study drug administration
3. Female using the following systemic contraceptives: oral, patch or vaginal ring, in the 28 days prior to the first study drug administration and during the study
4. Female using hormone replacement therapy in the 28 days prior to the first study drug administration and during the study
5. Female using the following systemic contraceptives: injections or implant, or hormone releasing intrauterine device in the 13 weeks prior to the first study drug administration and during the study
6. Drinking excessive amounts of tea, coffee, chocolate, and/or beverage or eating food containing caffeine (> 2 cups/day)
7. Use of tobacco or nicotine containing products (including but not limited to; cigarettes, electronic cigarettes, pipes, cigars, chewing tobacco, nicotine patch, or nicotine gum) within 90 days prior to the first study drug administration and the inability to abstain from nicotine containing products until the follow-up visit.
8. Past or current history of any mental, behavioral, or neurodevelopmental disorder as defined by the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) or significant risk of developing a psychosis (assessed by PRIME screen) or a personal history of psychotic symptoms (hallucinations or delusions) with or without a formal psychiatric diagnosis. Subjects with family history of significant mental, behavioral, or neurodevelopmental disorders unless determined by the Investigator (or designee) and agreed by the Medical Monitor to be non-clinically significant (NCS) will be excluded.
9. History or clinical manifestation of any metabolic, allergic, dermatological, hepatic, renal, hematological, pulmonary, gastrointestinal, neurological, respiratory, or endocrine disorder, unless determined by the Investigator (or designee) and agreed by the Medical Monitor to be NCS
10. Active or history of cardiovascular or cerebrovascular disease, including hypertension, angina, ischemic heart disease, transient ischemic attacks, bundle branch block, evidence of myocardial ischemia, stroke, and peripheral arterial disease sufficient to cause symptoms and/or require therapy to maintain stable status
11. History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, unless approved by the Investigator (or designee)
12. Active neoplastic disease or history of any neoplastic disease within 5 years of Screening (except for basal or squamous cell carcinoma of the skin or carcinoma in situ that has been definitely treated with standard of care)
13. Active infection (eg, sepsis, pneumonia, abscess) or a serious infection (eg, resulting in hospitalization or requiring parenteral antibiotic treatment) within 6 weeks prior to dosing
14. History of stomach or intestinal surgery or resection that would potentially alter absorption and/or excretion of orally administered drugs (uncomplicated appendectomy and hernia repair will be allowed)
15. Any of the following at Screening and/or prior to the first study drug administration:

    1. QT interval corrected for heart rate using Fridericia's method (QTcF) > 450 ms confirmed by repeat measurement
    2. QRS duration > 110 ms confirmed by confirmed by repeat measurement
    3. PR interval > 220 ms confirmed by repeat measurement
    4. Findings which would make QTc measurements difficult or QTc data uninterpretable
    5. History of additional risk factors for torsades de pointe (eg, heart failure, hypokalemia, family history of long QT syndrome)
16. Maintenance therapy with any drug or significant history of drug dependency or alcohol abuse (> 3 units of alcohol per day, intake of excessive alcohol, acute or chronic)
17. Positive test result for alcohol, cotinine, and/or drugs of abuse at Screening or prior to the first drug administration
18. Positive screening results to HIV Ag/Ab combo, hepatitis B surface antigen or hepatitis C virus tests
19. Any other clinically significant abnormalities in laboratory test results at Screening that would, in the opinion of an Investigator, increase the subject's risk of participation, jeopardize complete participation in the study, or compromise interpretation of study data
20. Intake of an IP in the 28 days prior to the first study drug administration
21. Use of any prescription drugs in the 28 days prior to the first study drug administration, that in the opinion of an Investigator would put into question the status of the participant as healthy
22. Use of St. John's wort in the 28 days prior to the first study drug administration and during the study
23. Consumption of any foods or beverages which alter CYP1A2 activity, e.g., barbecued food or cruciferous vegetables, such as broccoli and cauliflower, within 14 days prior to (first) check-in (a list of prohibited foods will be provided to subjects)
24. Consumption of any foods or beverages containing Seville-type oranges, grapefruit, or poppy seeds within 7 days prior to (first) check-in
25. Receipt of blood products within 2 months prior to check-in
26. Donation of 1 unit of blood to American Red Cross or equivalent organization or donation of over 500 mL of blood in the 56 days prior to the first study drug administration
27. Donation of plasma in the 7 days prior to the first study drug administration
28. Poor peripheral venous access
29. History or significant hypersensitivity to TMP301 or any related products (including excipients of the formulations) as well as severe hypersensitivity reactions (like angioedema) to any drugs
30. Subjects who, in the opinion of the Investigator (or designee; including input from subjects' general practitioner, as applicable), should not participate in this study
31. Subject hospitalized for any reason in a period of 30 days before the start of the study
32. Subjects who are investigational site staff members or directly involved in the conduct of the study and their family members or subjects who are employed by the Sponsor

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2023-01-06 (Actual); Primary Completion 2023-12-22 (Actual); Study Completion 2024-01-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dan Meyers, MD, Study Director — CMO, Tempero Bio
Locations (1):
- Altasciences, Overland Park, Kansas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1 - Active TMP-301: 50 mg BID Fasted
- Cohort 2 - Active TMP-301: 50 mg QD Fasted
- Cohort 3 - Active TMP-301: 50 mg QD Fed
- Cohort 4 - Active TMP-301: 25 mg QD Fed
Period: Overall Study
Arm/Group | Cohort 1 - Active TMP-301 | Cohort 2 - Active TMP-301 | Cohort 3 - Active TMP-301 | Cohort 4 - Active TMP-301 | Placebo
Started | 5 | 6 | 6 | 6 | 7
Completed | 0 | 5 | 5 | 5 | 6
Not Completed | 5 | 1 | 1 | 1 | 1
Not completed — Protocol-Specified Withdrawal | 5 | 0 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: 30
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 - Active TMP-301 | Cohort 2 - Active TMP-301 | Cohort 3 - Active TMP-301 | Cohort 4 - Active TMP-301 | Placebo | Total
Number analyzed (Participants) | 5 | 6 | 6 | 6 | 7 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.6 (8.17) | 47.8 (9.91) | 45.7 (10.42) | 32.0 (7.18) | 38.1 (8.51) | 40.1 (10.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 2 | 0 | 2 | 5
  Male | 5 | 5 | 4 | 6 | 5 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 0 | 0 | 1 | 3
  Not Hispanic or Latino | 4 | 4 | 6 | 6 | 6 | 26
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 1 | 2 | 2 | 3 | 10
  White | 3 | 3 | 3 | 4 | 3 | 16
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1 | 0 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 5 | 6 | 6 | 6 | 7 | 30

OUTCOME MEASURES:

1. Primary Outcome: Number of Treatment-Emergent Adverse Events (Safety and Tolerability)
Description: Occurence of Adverse Events, spontaneously reported and identified through clinical laboratory tests, vital sign measurements, ECG, physical exams and psychiatric assessments.
Time Frame: Within each cohort from screening to end of the follow up period up to 25 days
Measure: Number; unit: Number of TEAEs
Arm/Group | Cohort 1 - Active TMP-301 | Cohort 2 - Active TMP-301 | Cohort 3 - Active TMP-301 | Cohort 4 - Active TMP-301 | Placebo
Number analyzed (Participants) | 5 | 6 | 6 | 6 | 7
Number of TEAEs | 34 | 54 | 51 | 20 | 6

2. Secondary Outcome: To Evaluate the Plasma Area Under the Curve (AUC) 0-12 Hours After First Dose of TMP-301
Description: 0-12 hours post-dose on Day 1, twice daily dosing
Time Frame: Day 1
Population: Cohort 1 was twice daily dosing (BID). All other cohorts were once daily dosing (QD)
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Cohort 1 - Active TMP-301
Number analyzed (Participants) | 5
h*ng/mL | 888 (607)

3. Secondary Outcome: To Evaluate the Plasma Area Under the Curve (AUC) 0-24 Hours After First Dose of TMP-301
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Cohort 2 - Active TMP-301 | Cohort 3 - Active TMP-301 | Cohort 4 - Active TMP-301
Number analyzed (Participants) | 6 | 6 | 6
h*ng/mL | 1310 (848) | 1130 (345) | 489 (165)

4. Secondary Outcome: Maximum Plasma Concentration (Cmax) of TMP-301
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort 1 - Active TMP-301 | Cohort 2 - Active TMP-301 | Cohort 3 - Active TMP-301 | Cohort 4 - Active TMP-301
Number analyzed (Participants) | 5 | 6 | 6 | 6
ng/mL | 149 (86.5) | 224 (150) | 220 (93.9) | 97.5 (44.2)

5. Secondary Outcome: Time to Maximum Plasma Concentration (Tmax) of TMP-301
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Cohort 1 - Active TMP-301 | Cohort 2 - Active TMP-301 | Cohort 3 - Active TMP-301 | Cohort 4 - Active TMP-301
Number analyzed (Participants) | 5 | 6 | 6 | 6
h | 2.80 (0.84) | 2.67 (1.04) | 3.01 (1.11) | 3.17 (0.76)

6. Secondary Outcome: Plasma Concentration of TMP-301 at 12 Hours After First Dose (C12)
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort 1 - Active TMP-301 | Cohort 2 - Active TMP-301 | Cohort 3 - Active TMP-301 | Cohort 4 - Active TMP-301
Number analyzed (Participants) | 5 | 6 | 6 | 6
ng/mL | 33.3 (32.5) | 34.4 (25.4) | 23.2 (7.82) | 9.92 (4.43)

7. Secondary Outcome: Plasma Concentration of TMP-301 at 24 Hours After First Dose (C24)
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort 1 - Active TMP-301 | Cohort 2 - Active TMP-301 | Cohort 3 - Active TMP-301 | Cohort 4 - Active TMP-301
Number analyzed (Participants) | 5 | 6 | 6 | 6
ng/mL | 9.61 (17.2) | 9.23 (6.91) | 5.92 (1.56) | 2.32 (2.54)

8. Secondary Outcome: Maximum Plasma Concentration (Cmax) of TMP-301 at Steady State
Time Frame: Day 14
Population: Subjects in Cohort 1 were withdrawn after Day 8, therefore Day 14 pharmacokinetic parameters were not estimated for this cohort.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort 2 - Active TMP-301 | Cohort 3 - Active TMP-301 | Cohort 4 - Active TMP-301
Number analyzed (Participants) | 5 | 5 | 5
ng/mL | 464 (114) | 517 (125) | 220 (70.8)

9. Secondary Outcome: Average Plasma Concentration of TMP-301 at 12 Hours After Last Dose (C12)
Time Frame: Day 14
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort 2 - Active TMP-301 | Cohort 3 - Active TMP-301 | Cohort 4 - Active TMP-301
Number analyzed (Participants) | 5 | 5 | 5
ng/mL | 204 (50.3) | 193 (59.8) | 67.7 (21.0)

10. Secondary Outcome: Time to Maximum Plasma Concentration (Tmax) of TMP-301 at Steady State
Time Frame: Day 14
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Cohort 2 - Active TMP-301 | Cohort 3 - Active TMP-301 | Cohort 4 - Active TMP-301
Number analyzed (Participants) | 5 | 5 | 5
h | 1.86 (0.77) | 2.41 (1.13) | 2.41 (1.15)

11. Secondary Outcome: Minimum Drug Concentration (Cmin) of TMP-301 at Steady State
Time Frame: Day 14
Population: Subjects in Cohort 1 were withdrawn Day 8, therefore Day 14 pharmacokinetic parameters were not estimated for this cohort.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort 2 - Active TMP-301 | Cohort 3 - Active TMP-301 | Cohort 4 - Active TMP-301
Number analyzed (Participants) | 5 | 5 | 5
ng/mL | 125 (37.3) | 114 (44.7) | 30.1 (21.4)

12. Secondary Outcome: Area Under the Curve (Exposure) at Steady-state( AUC0_tau,ss), Over the Dosing Interval.
Time Frame: Day 14
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Cohort 2 - Active TMP-301 | Cohort 3 - Active TMP-301 | Cohort 4 - Active TMP-301
Number analyzed (Participants) | 5 | 5 | 5
h*ng/mL | 4910 (1210) | 4630 (1430) | 1630 (501)

13. Secondary Outcome: Plasma Concentration of TMP-301 at 24 Hours After Last Dose at Steady State (C24, ss)
Time Frame: Day 14
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort 2 - Active TMP-301 | Cohort 3 - Active TMP-301 | Cohort 4 - Active TMP-301
Number analyzed (Participants) | 5 | 5 | 5
ng/mL | 121 (27.9) | 120 (45.7) | 31.2 (20.6)

14. Secondary Outcome: Terminal Half-life (T1/2) of TMP-301
Time Frame: Day 14
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Cohort 2 - Active TMP-301 | Cohort 3 - Active TMP-301 | Cohort 4 - Active TMP-301
Number analyzed (Participants) | 5 | 5 | 5
h | 174.92 (139.78) | 125.86 (66.25) | 279.53 (378.19)

15. Secondary Outcome: Apparent Total Plasma Clearance of TMP-301 After Extravascular Administration (CL/F)
Time Frame: Day 14
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | Cohort 2 - Active TMP-301 | Cohort 3 - Active TMP-301 | Cohort 4 - Active TMP-301
Number analyzed (Participants) | 5 | 5 | 5
L/h | 10.7 (2.46) | 11.8 (4.10) | 16.4 (4.07)

16. Secondary Outcome: Apparent Volume of Distribution of TMP-301 at Steady State (Vz/F)
Time Frame: Day 14
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Cohort 2 - Active TMP-301 | Cohort 3 - Active TMP-301 | Cohort 4 - Active TMP-301
Number analyzed (Participants) | 5 | 5 | 5
L | 2610 (1930) | 2390 (1980) | 5010 (5010)

ADVERSE EVENTS:
Time Frame: 25 days
Arm/Group | Cohort 1 - Active TMP-301 | Cohort 2 - Active TMP-301 | Cohort 3 - Active TMP-301 | Cohort 4 - Active TMP-301 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/6 | 0/6 | 0/6 | 0/7
Serious Adverse Events (participants affected / at risk) | 1/5 | 0/6 | 0/6 | 0/6 | 0/7
Other Adverse Events (participants affected / at risk) | 4/5 | 6/6 | 6/6 | 2/6 | 2/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 - Active TMP-301 (N=5) | Cohort 2 - Active TMP-301 (N=6) | Cohort 3 - Active TMP-301 (N=6) | Cohort 4 - Active TMP-301 (N=6) | Placebo (N=7)
Worsening of psychotic disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 - Active TMP-301 (N=5) | Cohort 2 - Active TMP-301 (N=6) | Cohort 3 - Active TMP-301 (N=6) | Cohort 4 - Active TMP-301 (N=6) | Placebo (N=7)
Palpitations (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 2 | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 2 | 0 | 1 | 0 | 0
Asthenopia (Eye disorders) | 0 | 1 | 0 | 0 | 0
Diplopia (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0
Photophobia (Eye disorders) | 1 | 0 | 0 | 0 | 0
Rentinopathy solar (Eye disorders) | 1 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 1 | 0 | 0 | 0
Visual acuity reduced (Eye disorders) | 0 | 1 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Glossodynia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Paraesthesia oral (Gastrointestinal disorders) | 0 | 3 | 1 | 0 | 0
Feeling abnormal (General disorders) | 0 | 0 | 0 | 1 | 0
Feeling hot (General disorders) | 0 | 1 | 1 | 0 | 0
Feeling of relaxation (General disorders) | 0 | 0 | 1 | 1 | 0
Medical device site reaction (General disorders) | 0 | 3 | 0 | 1 | 0
Thirst (General disorders) | 0 | 0 | 1 | 0 | 0
Tinea cruris (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 2 | 0 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 0 | 1 | 0 | 0
Blood pressure increased (Investigations) | 1 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 0
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Balance disorder (Nervous system disorders) | 1 | 1 | 2 | 1 | 0
Disturbance in attention (Nervous system disorders) | 2 | 3 | 4 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 1 | 2 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 2 | 0 | 0 | 0
Headache (Nervous system disorders) | 2 | 4 | 3 | 0 | 1
Lethargy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Loss of proprioception (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 2 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 2 | 3 | 1 | 1
Tension headache (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Tremor (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Abnormal dreams (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Change in sustained attention (Psychiatric disorders) | 0 | 1 | 0 | 1 | 0
Depressed mood (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Derealisation (Psychiatric disorders) | 2 | 0 | 0 | 0 | 0
Euphoric mood (Psychiatric disorders) | 0 | 3 | 0 | 1 | 0
Hypervigilance (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Illusion (Psychiatric disorders) | 0 | 2 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 4 | 2 | 1 | 0 | 0
Intentional self-injury (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Irritability (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Libido decreased (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Psychotic disorder due to a general medical condition (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Tearfulness (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Time perception altered (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Peripheral coldness (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Ocular Dyscomfort (Eye disorders) | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator/site may not disclose, present, disseminate or produce any publication that contains information regarding the Services, Deliverables, or Study Data without Sponsor's prior written consent.

DOCUMENTS (2):
  • Study Protocol (2023-10-02): https://cdn.clinicaltrials.gov/large-docs/96/NCT06025396/Prot_000.pdf
  • Statistical Analysis Plan (2023-10-23): https://cdn.clinicaltrials.gov/large-docs/96/NCT06025396/SAP_001.pdf